CLINICAL TRIAL: NCT05315037
Title: Resistance Training Methods Impact On Glycemic Excursion and Metabolic Pathways in Type 1 Diabetes Mellitus
Brief Title: Resistance Training in Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Norton Healthcare (Other)
Responsible Party: Principal Investigator, Bradly Thrasher, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21.0565
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
Keywords: Resistance Training in type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Blood glucose and lactate measurements will be collected prior to any physical activity, post workout, and then 10- and 20-minutes post workout. Using a standard lancet device, capillary blood glucose values will be obtained using a Contour Next Glucometer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Training (Other): Bench press, Deadlift, Seated overhead press machine
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — Bench press: Exercise performed with participant lying supine with hands in prone position. Barbell is lowered vertically from fully extended elbow position to sternum, then returned to starting position. Barbell will be weighted with plates dependent on their strength and workout demands.
  Deadlift: Consists of gripping bar while in a squat position. Extension of ankles, knees, and hips while gripping the bar brings the weight up until joints are locked completing the exercise concentric portion. The eccentric lowering of the weight follows and consists of flexion of joints.
  Seated overhead press machine: This multi-joint exercise, deltoid and trapezius are the prime movers and triceps are secondary movers, with hands on the grips and a position allowing back and buttocks to be completely supported. They push against a load vertically until glenohumeral joint fully extends, then load is returned to starting position and process continues until all repetitions desired are achieved

SUMMARY:
The purpose of this study is to learn how different resistance training programs affects blood sugar in young athletes with T1DM.

DETAILED DESCRIPTION:
Strength and condition training to improve sport performance has been greatly emphasized over the past 20 years. Formal strength and conditioning (S&C) programming is performed by S&C coaches who are educated in the field of exercise program with the intentions to bring about particular athletic adaptations through exercise. S&C programs, previously limited to programs at the college and professional level, are now commonly seen in secondary school athletic programs. With such broad adoption, many athletes that manage chronic diseases, such as type 1 diabetes mellitus, are exposed to elements of these programs.

Diabetes mellitus impacts more than 10% of the United States population. Of these, 5.2% have identified type 1 diabetes mellitus (T1DM) which includes approximately 210,000 individuals under the age of 20. In addition to insulin and dietary management, exercise and physical activity is recommended as an important therapeutic tool for most patients with T1DM. Physical activity has been shown to significantly improve glycemic control in individuals with diabetes. Additional benefits of exercise include improved cardiovascular fitness, muscle strength, insulin sensitivity and blood glucose control. S&C programs offer benefits to those living with T1DM as different exercises can be tailored to preserve health. However, there are no exercise prescription or guidelines specifically for adolescent athletes diagnosed with type 1 diabetes participating in strength and conditioning programs. Furthermore, there is no available data that states the predictability of glucose response and insulin needs to any of the specific strength and conditioning goals.

Objective: To assess the impact of different strength and conditioning programming on glycemic control in athletes with T1DM.

Primary Aim: Assess glucose response to different resistance training methods. Secondary Aims: To assess for correlation between lactate and glucose using different resistance training methods.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 13 years of age
* ≥2 years from date of T1DM diagnosis
* Prior exposure to strength and conditioning
* HbA1C ≤ 10%
* Actively utilizing continuous glucose monitoring for diabetes management

Exclusion Criteria:

* Physical limitation that may impede ability to complete study procedures
* Non-English-speaking individual

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess glucose response to different resistance training methods | 3 months
  Blood glucose

SECONDARY OUTCOMES:
To assess for correlation between lactate and glucose using different resistance training methods | 3 months
  Blood glucose, lactate

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No